CLINICAL TRIAL: NCT04140422
Title: Efficacy of Hyperosmolar Eye Drops in Diurnal Corneal Edema in Fuchs Endothelial Dystrophy: a Double Blind Randomized Controlled Trial
Brief Title: Eye Drops for Early Morning-Associated Corneal Swelling of the Cornea
Acronym: EDEMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Eye Hospital, Freiburg (Other)
Responsible Party: Principal Investigator, Katrin Wacker, MD, Principal Investigator, University Eye Hospital, Freiburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETK 366/19
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Fuchs' Endothelial Dystrophy
Keywords: Corneal edema; Descemet membrane endothelial keratoplasty (DMEK); Hyperosmolar eye drops
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Corneal Edema

STUDY DESIGN:
Intervention Model Description: The study uses both eyes of the participant to allow inter- and intraindividual comparisons. One eye will be randomized to be treated with hyperosmolar eye drops, the fellow eye will be treated with lubricating eye drops.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The allocation is done randomly by the hospitals pharmacy. By using identical containers for the hyperosmolar eye drops and the lubricating eye drops participants and medical staff are not able to distinguish both substances.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperosmolar Eye Drops (Experimental): 5% sodium chloride eye drops with 0,15% hyaluronic acid; one drop after waking up and one drop 30 min later on study day; investigator administered
  Interventions: Other: Hyperosmolar eye drops
- Lubricating Eye Drops (Placebo Comparator): Lubricating eye drops with 0,15% hyaluronic acid; one drop after waking up and one drop 30 min later on study day; investigator administered
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Hyperosmolar eye drops — Application of one preservative-free hyperosmolar eye drop, when waking up and one eye drop 30 min later to one eye by the investigators
  Other Names: ODM 5 (CE0459)
  Arms: Hyperosmolar Eye Drops
Other: Placebo — Application of one preservative-free lubricating eye drop, when waking up and one eye drop 30 min later to the fellow eye by the investigators
  Other Names: Placebo (for hyperosmolar eye drops)
  Arms: Lubricating Eye Drops

SUMMARY:
This study evaluates the efficacy of hyperosmolar eye drops on early morning edema of the cornea in patients with Fuchs' endothelial corneal dystrophy (FECD). Each participant will receive hyperosmolar eye drops in one eye and lubricating eye drops in the fellow eye.

DETAILED DESCRIPTION:
Hyperosmolar eye drops are lubricating eye drops with 5% of sodium chloride. Hyperosmolar eye drops are thought to temporarily deswell the cornea.

During morning hours, patients with Fuchs' endothelial corneal dystrophy (FECD) typically report poor vision and disturbing glare because of corneal edema. To improve vision in advanced stages of the disease, corneal endothelial transplantation has become the treatment of choice. Many patients with Fuchs' endothelial corneal dystrophy (FECD) use hyperosmolar eye drops before transplantation. At present, it is unclear, how much hyperosmolar eye drops help reducing corneal edema in Fuchs' endothelial corneal dystrophy (FECD). Based on our previous work that determined the amount of additional corneal edema in the morning in patients with Fuchs' endothelial corneal dystrophy (FECD), the investigators will assess if hyperosmolar eye drops speed up the deswelling process.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced Fuchs' endothelial corneal dystrophy (FECD)
* Indication for corneal endothelial transplantation (Descemet Membrane Endothelial Keratoplasty - DMEK)
* Must be able to speak and understand German or English.

Exclusion Criteria:

* Other corneal diseases (i.e. epithelial defects except for bullae caused by Fuchs' endothelial corneal dystrophy (FECD), corneal scars, postoperative / bullous keratopathy, corneal degenerations / dystrophies, corneal inflammation / infection)
* Regular use of drugs potentially affecting the cornea (i.e. amiodarone, chloroquine, triptan, isotretinoin, constant use of antihistamines, use of contact lenses in past four weeks, anesthetic eye drops, corticosteroid eye drops, antibiotic eye drops in past four weeks, glaucoma drops, hyperosmolar eye drops within the past 24 hours)
* Systemic diseases that affect the cornea (e.g. connective tissue disease, complicated diabetes mellitus)
* Lack of fixation during corneal tomography

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Change in corneal thickness | Between eye opening in the morning (7 am; Hour 0) and 1 hour later (Hour 1)
  Tomography to determine the thickness of the cornea

SECONDARY OUTCOMES:
Change in corneal thickness over time | Over the first 4 hours after eye opening (Hour 0 to Hour 4) and at presumed steady-state in the afternoon (Hour 9)
  Tomography to determine the thickness of the cornea
Change in corneal backscatter over time | Over the first 4 hours after eye opening (Hour 0 to Hour 4) and at presumed steady-state in the afternoon (Hour 9)
  Tomography to determine corneal backscatter
Change in forward scatter over time | Over the first 4 hours after eye opening (Hour 0 to Hour 4) and at presumed steady-state in the afternoon (Hour 9)
  Stray light meter measurement to determine the forward scatter
Change in visual acuity over time | Over the first 4 hours after eye opening (Hour 0 to Hour 4) and at presumed steady-state in the afternoon (Hour 9)
  Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity charts to determine visual acuity
Change in subjective visual acuity | Over the first 4 hours after eye opening (Hour 0 to Hour 4) and at presumed steady-state in the afternoon (Hour 9)
  Question on presumed change of vision

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Wacker, MD, Principal Investigator — University of Freiburg, Eye Hospital
Locations (1):
- Medical Center - University of Freiburg, Eye Hospital, Freiburg im Breisgau, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fritz M, Grewing V, Maier P, Lapp T, Bohringer D, Reinhard T, Wacker K. Diurnal Variation in Corneal Edema in Fuchs Endothelial Corneal Dystrophy. Am J Ophthalmol. 2019 Nov;207:351-355. doi: 10.1016/j.ajo.2019.08.002. Epub 2019 Aug 12. PMID 31415734
- [Background] Wacker K, Baratz KH, Bourne WM, Patel SV. Patient-Reported Visual Disability in Fuchs' Endothelial Corneal Dystrophy Measured by the Visual Function and Corneal Health Status Instrument. Ophthalmology. 2018 Dec;125(12):1854-1861. doi: 10.1016/j.ophtha.2018.06.018. Epub 2018 Aug 10. PMID 30104038
- [Background] Wilson SE, Bourne WM. Fuchs' dystrophy. Cornea. 1988;7(1):2-18. PMID 3280235
- [Derived] Zander DB, Bohringer D, Fritz M, Grewing V, Maier PC, Lapp T, Reinhard T, Wacker K. Hyperosmolar Eye Drops for Diurnal Corneal Edema in Fuchs' Endothelial Dystrophy: A Double-Masked, Randomized Controlled Trial. Ophthalmology. 2021 Nov;128(11):1527-1533. doi: 10.1016/j.ophtha.2021.04.015. Epub 2021 Apr 20. PMID 33892048